CLINICAL TRIAL: NCT06375070
Title: Anticoagulants for PFO Patients
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: RMeng1
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Patent Foramen Ovale
Keywords: patent foramen ovale; migraine; stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders; Stroke | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- small-shunt Group: small (3-9 bubbles)
  Interventions: Procedure: PFO closure; Drug: anticoagulant
- moderate-shunt Group: (10-30 bubbles)
  Interventions: Procedure: PFO closure; Drug: anticoagulant
- large-shunt Group: >30 bubbles
  Interventions: Procedure: PFO closure; Drug: anticoagulant

INTERVENTIONS:
Procedure: PFO closure — PFO closure
Drug: anticoagulant — rivaroxaban

SUMMARY:
Patients who underwent both bubble transcranial Doppler (bubble-TCD) and transoesophageal echocardiography (TEE) at our institution were consecutively enrolled in this real-world case-control study from August 2016 through August 2023. The patients were categorized into three groups based on the degree of the shunt observed: mild (3-9 bubbles), moderate (10-30bubbles), and severe (more than 30 bubbles). In cases with mild-shunt (small-size) PFO, post-procedural anticoagulation or PFO closure was administered. Subsequent to the interventions, the follow-up encompassed the recording of migraine remission, recurrent neurological incidents, instances of major bleeding, and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. verified PFO diagnosis through TEE, Bubble-TCD, or contrast echocardiography of the right heart;
2. ages range between 16 and 65;
3. no restrictions on sexual orientation;
4. stroke patients with cryptogenic strokes as per the TOAST classification;
5. no other likely causes for migraines, with the exception of PFO;
6. no multiple risk factors for cerebrovascular disease, such as hypertension, diabetes, or smoking.

Exclusion Criteria:

* 1)severe, acute, or life-threatening conditions including acute cardio-cerebrovascular diseases, significant organ failure, or infections; 2)magnetic resonance imaging (MRI) contraindications, especially with contrast enhancement; 3) presence of cerebral artery stenosis, internal carotid artery stenosis, or atherosclerosis; 4) hypercoagulability or venous thrombosis; 5) contraindications associated with PFO closure and anticoagulants; 6) obstructive sleep apnea.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants had their PFO diagnosis confirmed via transoesophageal echocardiography (TEE), bubble transcranial Doppler (Bubble-TCD), or contrast echocardiography of the right heart and gave their informed consent to participate
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
whether occur recurrent stroke or migraine relief | 12 months

IPD SHARING:
Plan to Share IPD: No